CLINICAL TRIAL: NCT05623709
Title: Health Outcomes Following Treatment With Continuous Positive Airway Pressure or Noninvasive Ventilation in Patients With Chronic Obstructive Pulmonary Disease and a Sleep Related Breathing Disorder
Brief Title: Health Outcomes With CPAP or NIV in Patients With COPD and a Sleep Related Breathing Disorder
Status: Terminated | Type: Observational
Why Stopped: Recruitment difficulties
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00118055
Record Dates: First submitted 2022-11-11; First posted 2022-11-21 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Sleep Related Hypoventilation; Obstructive Sleep Apnea; Hypoventilation
Keywords: continuous positive airway pressure; bilevel positive airway pressure; noninvasive ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive; Hypoventilation | interventions — Continuous Positive Airway Pressure; Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- COPD and SRBD prescribed NIV or CPAP: Group 1a: (n=55) Adults with a SRBD and COPD who are newly prescribed NIV treatment within the study period.
  Group 1b: (n=55) Adults with a SRBD and COPD who are newly prescribed CPAP treatment within the study period.
  Interventions: Device: Positive airway pressure with continuous positive airway pressure or noninvasive ventilation
- COPD controls not prescribed CPAP or NIV: Group 2: COPD controls without a SRBD: (n=55) Adults with COPD who undergo sleep diagnostic testing and who are not recommended to start CPAP or NIV

INTERVENTIONS:
Device: Positive airway pressure with continuous positive airway pressure or noninvasive ventilation — CPAP or NIV prescribed by the treating respirologist for long-term use at home
  Other Names: CPAP, NIV, PAP treatment
  Groups: COPD and SRBD prescribed NIV or CPAP

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic lung disease affecting an estimated 1 in 10 Canadians. Symptoms include persistent shortness of breath, cough and sputum production. The symptoms can be serious when people with COPD experience a flare of their disease and may lead to hospitalization or death. Improving other conditions that affect COPD control is one way to improve the health of people with COPD. Obstructive sleep apnea (OSA) is the most common breathing problem during sleep, and commonly co-exists with COPD. Although diagnosing and treating OSA is encouraged, it has not been highlighted in guidelines that recommend ideal COPD care. People with COPD and OSA have lower sleep quality and lower oxygen levels during sleep compared to people with OSA. Despite these differences, treatment of OSA in people with COPD is modeled after treatment of OSA in the general population, generally using treatment with continuous positive airway pressure (CPAP) with the possible addition of oxygen through the CPAP machine. There are few studies looking at other types of treatment including noninvasive ventilation (NIV) in people with COPD and OSA. The majority of studies of NIV in COPD has been for people with other reasons to use NIV including acute respiratory failure or chronic hypercarbic respiratory failure and did not include people with risk factors for OSA or who had undergone overnight sleep studies.

In Alberta, NIV is provided province wide for people who have both OSA who do not meet certain physiologic targets in their oxygen levels or breathing patterns after CPAP is applied on an overnight sleep study. NIV is provided preferentially to CPAP and oxygen, providing an opportunity to look at health outcomes when NIV is used instead of CPAP for the treatment of patients with COPD. Through this study, we will measure whether people with COPD and a sleep related breathing disorder such as OSA have fewer severe flares of COPD after starting CPAP or NIV. We will evaluate whether the number of Emergency Department visits, hospitalizations or deaths lowers after starting CPAP or NIV.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease is a common chronic lung disease affecting more than 10% of Canadians. Patients with COPD have significant morbidity from the disease as almost 60% of Albertans living with COPD were hospitalized between 2012-2014. Sleep related breathing disorders (SRBD) are a common comorbidity of COPD, and contribute to the morbidity associated with COPD. The most common SRBD is OSA. It is estimated that 1.0-3.6% of Canadians are affected by both OSA and COPD. People with COPD and OSA have lower sleep quality, lower oxygen saturations and greater nocturnal oxygen desaturations when their sleep is compared to people with OSA. Observational studies suggest that patients with OSA and COPD have a higher risk of hospitalization, exacerbation of COPD, or death; however, the evidence to support the assessment and management of OSA improving COPD health outcomes has not been considered substantial enough to justify inclusion in COPD guidelines. Other SRBDs that may impact patients with COPD are sleep-related hypoventilation as a consequence of obesity, or central sleep apnea as a consequence of cardiac disease, stroke or use of opioids; however, these are less common and less studied types of SRBD within sleep literature.

Two treatments that are commonly prescribed for SRBD are CPAP or NIV. In patients with OSA, CPAP improves quality of life, daytime sleepiness, and blood pressure control. In patients with COPD who have OSA, observational studies suggest that CPAP use is associated with survival, with the duration of CPAP use per night lowering mortality in a dose dependent manner, an increased time to first moderate-severe COPD exacerbation and fewer hospitalizations related to exacerbations of COPD. The association of decreased health care utilization with CPAP is greater in patients with a higher COPD complexity and number of comorbidities, indicating those who are the sickest may derive the most harm from untreated disease. NIV is better tolerated than CPAP in some patients with OSA; yet, there have been only a few studies evaluating its use for a SRBD in COPD. Further work in this area is critically important as the indications for use of NIV are expanding among patients with COPD.

We are uniquely positioned to complete this study as NIV is provided province-wide in Alberta and patient health outcomes are available in provincial databases. In addition, within the provincial titration protocol for polysomnography, NIV is provided preferentially over CPAP with oxygen, differentiating the management of these patients from the titration protocols used in other studies.

Through this study, we will explore whether treatment with NIV or CPAP for a SRBD in patients with COPD results in fewer moderate-severe exacerbations of COPD and whether the use of these devices have an impact on health care utilization and mortality. In a subgroup analysis, we will explore whether NIV use results in similar outcomes as CPAP, and account for differences in disease severity in this comparison. Adherence with these CPAP or NIV will also be summarized. The results from this study will inform regional care as well as provide insight into the roles of CPAP and NIV in the treatment of SRBD in patients with COPD.

Sample size:

59% of Albertans with COPD experience an exacerbation within a 2 year period; however, a conservative estimate of 50% will be used for the power calculation. A clinically significant difference in COPD exacerbations is estimated to be 25%. An estimated standard deviation of 8 patients hospitalized per 2 years was estimated (variance 64). Given that the exposure group will be stratified by use of CPAP or NIV in subgroup analysis, a 2:1 proportion for the exposure to comparison group was utilized and the exposure arm will be composed of equal proportions of patients prescribed CPAP or NIV. A 10% drop out rate is anticipated.

Primary hypothesis: Null hypothesis (H0): CPAP or NIV is equivalent to no therapy; Alternate hypothesis (H1): CPAP or NIV is better than no therapy

Secondary hypothesis: Null hypothesis (H0): NIV is equivalent to CPAP; Alternate hypothesis (H1): NIV is better than CPAP

For the primary hypothesis, these estimates suggest that a sample size of 165 patients is required (n=110 patients in the exposure arm and 55 patients in the control arm). For the secondary hypothesis, it is not anticipated that a large difference between CPAP or NIV will be observed; however, the subgroup analysis of the primary outcome will be powered to detect a 25% difference between intervention with CPAP or NIV.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults who have completed polysomnography at the University of Alberta Sleep Disorders Laboratory in Edmonton, Alberta, Canada.
* Naïve to CPAP or NIV therapy or have use of CPAP or NIV <4 weeks in the past
* Diagnosed with COPD by a respirologist and has fixed airflow obstruction on spirometry (i.e., post-bronchodilator FEV1/FVC <LLN on spirometry or FEV1/FVC <0.70 if the LLN is not provided)
* Diagnosed with a SRBD for which CPAP or NIV are commonly prescribed, as defined below; some of the patients with mild SRBD or a SRBD suspected to be secondary to COPD rather than OSA (e.g. mild OSA, sustained hypercarbia, hypoxemia etc) may not be prescribed CPAP or NIV at the treating physician's discretion

  * OSA will be defined as a predominantly obstructive apnea-hypopnea index (AHI) ≥5 events/hr of sleep on sleep diagnostic testing in the presence of symptoms/relevant comorbidities or an AHI ≥15 events/hr irrespective of symptoms. If home sleep apnea testing was used in place of polysomnography, the respiratory event index (REI) will be a surrogate of AHI.
  * Hypoventilation will be defined by polysomnography criteria as a sustained elevation in the TcCO2 to be >55 mmHg for ≥10 min or a rise in TcCO2 by >10 mmHg to a value >50 mmHg for ≥10 min. If an arterial blood gas is available, sustained hypercapnia as defined by arterial carbon dioxide oxygen tension (PaCO2) >45 mmHg or serum bicarbonate (HCO3) ≥27 mmol/L while medically stable will be reported.

Exclusion Criteria:

* Significant lung disease in addition to COPD
* Neuromuscular disease including diaphragmatic paralysis
* Dementia
* Treatment with CPAP or NIV for >4 weeks prior to study eligibility.
* Refusal to participate
* Inability to consent in English and do not have an interpreter readily available
* Current diagnosis of an active malignancy
* Central sleep apnea as the indication for PAP treatment. Central sleep apnea will be defined as a central hypopnea index ≥5 events/hr of sleep on polysomnography and the number of central apneas and/or central hypopneas is >50% of the AHI with or without Cheyne-Stokes breathing

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study setting are people living in Alberta receiving care by an adult respirologist who undergo sleep diagnostic testing, consent to contact for research at a participating site, are eligible for the study after a brief chart review, and who subsequently consent to be involved in the study. The start date for CPAP or NIV will need to be within the study period although it will not need to be after the date of sleep diagnostic testing in order to allow patients started on NIV in hospital who subsequently undergo sleep diagnostic testing to be eligible. Polysomnograms for eligible patients will be completed by sleep laboratories operating within Alberta Health Services within the public health care system. Home sleep apnea tests are performed by both private and public facilities within Alberta and both sites of testing will be considered adequate for patient inclusion in the study if that is the sole form of sleep diagnostic testing requested by the treating respirologist.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with moderate-severe exacerbations of COPD (Emergency Department visit for COPD) in the 2 years following initiation of CPAP or NIV compared to the 2 years prior | 2 years
  [stratified by intervention with CPAP or NIV]

SECONDARY OUTCOMES:
Proportion of patients with severe exacerbation of COPD (hospitalization/intensive care unit admission for COPD) in the 2 years following initiation of CPAP or NIV compared to the 2 years prior | 2 years
  [stratified by intervention with CPAP or NIV]
Mean difference in the number of days hospitalized in the 2 years after the date of CPAP or NIV initiation or date of sleep diagnostic testing compared to the 2 years prior | 2 years
  [stratified by intervention with CPAP or NIV] [stratified by all-cause, stroke, cardiovascular, exacerbation of COPD or respiratory cause] Total number of days hospitalized [stratified by number of events/year]
Mean difference in hospitalizations/intensive care unit admissions for severe exacerbations of COPD in the 2 years after the date of CPAP or NIV initiation or date of sleep diagnostic testing compared to the 2 years prior | 2 years
  [stratified by intervention with CPAP or NIV] Number of events [stratified by number of events/year] Time to event
Mean difference in Emergency Department visits for moderate-severe exacerbations of COPD in the 2 years after the date of CPAP or NIV initiation or date of sleep diagnostic testing compared to the 2 years prior | 2 years
  [stratified by intervention with CPAP or NIV] Number of events [stratified by number of events/year] Time to event
Composite outcome of Emergency Department visits or hospitalizations following the date of NIV or CPAP initiation or date of sleep diagnostic testing | 2 years
  [stratified by all-cause, stroke, cardiovascular, exacerbation of COPD or respiratory cause] [stratified by intervention with CPAP or NIV]
Mortality following the start of NIV or CPAP or following the date of sleep diagnostic testing | 2 years
  [stratified by all-cause, stroke, cardiovascular, exacerbation of COPD or respiratory cause] [stratified by intervention with CPAP or NIV]
Mean and median hours of use of CPAP or NIV in hours/day | 2 years
  [Stratified by intervention with CPAP or NIV]

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Given that this is a phase IV clinical trial, the information will be disseminated through publication. Requests for IPD data from this study will need to go through institutional ethics review prior to use for a secondary purpose.

REFERENCES:
- [Background] Shawon MS, Perret JL, Senaratna CV, Lodge C, Hamilton GS, Dharmage SC. Current evidence on prevalence and clinical outcomes of co-morbid obstructive sleep apnea and chronic obstructive pulmonary disease: A systematic review. Sleep Med Rev. 2017 Apr;32:58-68. doi: 10.1016/j.smrv.2016.02.007. Epub 2016 Mar 2. PMID 28169105
- [Background] Donovan LM, Feemster LC, Udris EM, Griffith MF, Spece LJ, Palen BN, He K, Parthasarathy S, Strohl KP, Kapur VK, Au DH. Poor Outcomes Among Patients With Chronic Obstructive Pulmonary Disease With Higher Risk for Undiagnosed Obstructive Sleep Apnea in the LOTT Cohort. J Clin Sleep Med. 2019 Jan 15;15(1):71-77. doi: 10.5664/jcsm.7574. PMID 30621828
- [Background] Marin JM, Soriano JB, Carrizo SJ, Boldova A, Celli BR. Outcomes in patients with chronic obstructive pulmonary disease and obstructive sleep apnea: the overlap syndrome. Am J Respir Crit Care Med. 2010 Aug 1;182(3):325-31. doi: 10.1164/rccm.200912-1869OC. Epub 2010 Apr 8. PMID 20378728
- [Background] Criner GJ, Bourbeau J, Diekemper RL, Ouellette DR, Goodridge D, Hernandez P, Curren K, Balter MS, Bhutani M, Camp PG, Celli BR, Dechman G, Dransfield MT, Fiel SB, Foreman MG, Hanania NA, Ireland BK, Marchetti N, Marciniuk DD, Mularski RA, Ornelas J, Road JD, Stickland MK. Prevention of acute exacerbations of COPD: American College of Chest Physicians and Canadian Thoracic Society Guideline. Chest. 2015 Apr;147(4):894-942. doi: 10.1378/chest.14-1676. PMID 25321320
- [Background] O'Donnell DE, Aaron S, Bourbeau J, Hernandez P, Marciniuk D, Balter M, Ford G, Gervais A, Goldstein R, Hodder R, Maltais F, Road J; Canadian Thoracic Society. Canadian Thoracic Society recommendations for management of chronic obstructive pulmonary disease--2003. Can Respir J. 2003 May-Jun;10 Suppl A:11A-65A. doi: 10.1155/2003/567598. English, French. PMID 12861361
- [Background] Laratta CR, Ayas NT, Povitz M, Pendharkar SR. Diagnosis and treatment of obstructive sleep apnea in adults. CMAJ. 2017 Dec 4;189(48):E1481-E1488. doi: 10.1503/cmaj.170296. No abstract available. PMID 29203617
- [Background] Machado MC, Vollmer WM, Togeiro SM, Bilderback AL, Oliveira MV, Leitao FS, Queiroga F Jr, Lorenzi-Filho G, Krishnan JA. CPAP and survival in moderate-to-severe obstructive sleep apnoea syndrome and hypoxaemic COPD. Eur Respir J. 2010 Jan;35(1):132-7. doi: 10.1183/09031936.00192008. Epub 2009 Jul 2. PMID 19574323
- [Background] Stanchina ML, Welicky LM, Donat W, Lee D, Corrao W, Malhotra A. Impact of CPAP use and age on mortality in patients with combined COPD and obstructive sleep apnea: the overlap syndrome. J Clin Sleep Med. 2013 Aug 15;9(8):767-72. doi: 10.5664/jcsm.2916. PMID 23946706
- [Background] Singh G, Agarwal A, Zhang W, Kuo YF, Sultana R, Sharma G. Impact of PAP therapy on hospitalization rates in Medicare beneficiaries with COPD and coexisting OSA. Sleep Breath. 2019 Mar;23(1):193-200. doi: 10.1007/s11325-018-1680-0. Epub 2018 Jun 22. PMID 29931497
- [Background] Kaminska M, Rimmer KP, McKim DA, Nonoyama M, Giannouli E, Morrison Debra L, et al. Long-term non-invasive ventilation in patients with chronic obstructive pulmonary disease (COPD): 2021 Canadian Thoracic Society Clinical Practice Guideline update. Canadian Journal of Respiratory, Critical Care, and Sleep Medicine. 2021;5(3):160-83.
- [Background] Leung C, Bourbeau J, Sin DD, Aaron SD, FitzGerald JM, Maltais F, Marciniuk DD, O'Donnell D, Hernandez P, Chapman KR, Walker B, Road JD, Zheng L, Zou C, Hogg JC, Tan WC; CanCOLD Collaborative Research Group. The Prevalence of Chronic Obstructive Pulmonary Disease (COPD) and the Heterogeneity of Risk Factors in the Canadian Population: Results from the Canadian Obstructive Lung Disease (COLD) Study. Int J Chron Obstruct Pulmon Dis. 2021 Feb 12;16:305-320. doi: 10.2147/COPD.S285338. eCollection 2021. PMID 33603357
- [Background] Canadian Institute for Health Information. COPD in Alberta: Examining the Characteristics and Health Care Use of High Users. Ottawa, ON: CIHI; 2017.
- [Background] Ishak A, Ramsay M, Hart N, Steier J. BPAP is an effective second-line therapy for obese patients with OSA failing regular CPAP: A prospective observational cohort study. Respirology. 2020 Apr;25(4):443-448. doi: 10.1111/resp.13674. Epub 2019 Aug 12. PMID 31407464
- [Background] Murphy PB, Arbane G, Ramsay M, Suh ES, Mandal S, Jayaram D, Leaver S, Polkey MI, Hart N. Safety and efficacy of auto-titrating noninvasive ventilation in COPD and obstructive sleep apnoea overlap syndrome. Eur Respir J. 2015 Aug;46(2):548-51. doi: 10.1183/09031936.00205714. Epub 2015 Jun 25. No abstract available. PMID 26113686
- [Background] Duiverman ML, Wijkstra PJ. Long-Term Noninvasive Ventilation in COPD: Is High-Intensity NIV The Way To Go? Chronic Obstr Pulm Dis. 2015 Dec 14;3(1):378-381. doi: 10.15326/jcopdf.3.1.2015.0179. No abstract available. PMID 28848859
- [Background] Macrea M, Oczkowski S, Rochwerg B, Branson RD, Celli B, Coleman JM 3rd, Hess DR, Knight SL, Ohar JA, Orr JE, Piper AJ, Punjabi NM, Rahangdale S, Wijkstra PJ, Yim-Yeh S, Drummond MB, Owens RL. Long-Term Noninvasive Ventilation in Chronic Stable Hypercapnic Chronic Obstructive Pulmonary Disease. An Official American Thoracic Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2020 Aug 15;202(4):e74-e87. doi: 10.1164/rccm.202006-2382ST. PMID 32795139
- [Background] Ergan B, Oczkowski S, Rochwerg B, Carlucci A, Chatwin M, Clini E, Elliott M, Gonzalez-Bermejo J, Hart N, Lujan M, Nasilowski J, Nava S, Pepin JL, Pisani L, Storre JH, Wijkstra P, Tonia T, Boyd J, Scala R, Windisch W. European Respiratory Society guidelines on long-term home non-invasive ventilation for management of COPD. Eur Respir J. 2019 Sep 28;54(3):1901003. doi: 10.1183/13993003.01003-2019. Print 2019 Sep. PMID 31467119
- [Background] American Academy of Sleep Medicine. International classification of sleep disorders, 3rd ed. Darien. IL: American Academy of Sleep Medicine, 2014.
- [Background] Berry RB, Brooks R, Gamaldo CE, et al. The AASM manual for the scoring of sleep and associated events: rules, terminology and technical specifications, version 2.3. Darien (II): American Academy of Sleep Medicine; 2016.
- [Background] Randerath W, Verbraecken J, Andreas S, Arzt M, Bloch KE, Brack T, Buyse B, De Backer W, Eckert DJ, Grote L, Hagmeyer L, Hedner J, Jennum P, La Rovere MT, Miltz C, McNicholas WT, Montserrat J, Naughton M, Pepin JL, Pevernagie D, Sanner B, Testelmans D, Tonia T, Vrijsen B, Wijkstra P, Levy P. Definition, discrimination, diagnosis and treatment of central breathing disturbances during sleep. Eur Respir J. 2017 Jan 18;49(1):1600959. doi: 10.1183/13993003.00959-2016. Print 2017 Jan. PMID 27920092
- [Background] Chapman KR, Bergeron C, Bhutani M, Bourbeau J, Grossman RF, Hernandez P, McIvor RA, Mayers I. Do we know the minimal clinically important difference (MCID) for COPD exacerbations? COPD. 2013 Apr;10(2):243-9. doi: 10.3109/15412555.2012.733463. Epub 2013 Mar 20. PMID 23514218
- [Background] Ballard RD, Gay PC, Strollo PJ. Interventions to improve compliance in sleep apnea patients previously non-compliant with continuous positive airway pressure. J Clin Sleep Med. 2007 Dec 15;3(7):706-12. PMID 18198804
- [Background] Fleetham J, Ayas N, Bradley D, Ferguson K, Fitzpatrick M, George C, Hanly P, Hill F, Kimoff J, Kryger M, Morrison D, Series F, Tsai W; CTS Sleep Disordered Breathing Committee. Canadian Thoracic Society guidelines: diagnosis and treatment of sleep disordered breathing in adults. Can Respir J. 2006 Oct;13(7):387-92. doi: 10.1155/2006/627096. No abstract available. PMID 17036094